CLINICAL TRIAL: NCT06012240
Title: A Phase 3 Randomized, Placebo-controlled, Double-blind Program to Evaluate Efficacy and Safety of Upadacitinib in Adult and Adolescent Subjects With Severe Alopecia Areata
Brief Title: A Study to Evaluate the Safety and Effectiveness of Upadacitinib Tablets in Adult and Adolescent Participants With Severe Alopecia Areata
Acronym: Up-AA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M23-716; 2023-505061-82-01 (Other: EU CT)
Record Dates: First submitted 2023-08-22; First posted 2023-08-25 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Alopecia Areata
Keywords: Alopecia Areata; Upadacitinib; Rinvoq; ABT-494
MeSH Terms: conditions — Alopecia Areata | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (23):
- Study 1: Group 1 Upadacitinib Dose A (Experimental): Participants will receive upadacitinib Dose A once daily for 52 weeks in Period A and Period B.
  Interventions: Drug: Upadacitinib
- Study 1: Group 2 Upadacitinib Dose B (Experimental): Participants will receive upadacitinib Dose B once daily for 52 weeks in Period A and Period B.
  Interventions: Drug: Upadacitinib
- Study 1: Group 3 Placebo (Experimental): Participants will receive matching placebo once daily for 24 weeks in Period A.
  Interventions: Drug: Placebo
- Study 1: Group 4 Upadacitinib Dose A (Experimental): Participants initially randomized to placebo (Period A) with a SALT score > 20 at Week 24 will be re-randomized to receive upadacitinib Dose A once daily for 28 weeks in Period B.
  Interventions: Drug: Upadacitinib; Drug: Placebo
- Study 1: Group 5 Upadacitinib Dose B (Experimental): Participants initially randomized to placebo (Period A) with a SALT score > 20 at Week 24 will be re-randomized to receive upadacitinib Dose B once daily for 28 weeks in Period B.
  Interventions: Drug: Upadacitinib; Drug: Placebo
- Study 1: Group 6 Placebo (Experimental): Participants initially randomized to placebo with a SALT score ≤ 20 at Week 24 will continue on placebo through Week 160.
  Interventions: Drug: Placebo
- Study 2: Group 1 Upadacitinib Dose A (Experimental): Participants will receive upadacitinib Dose A once daily for 52 weeks in Period A and Period B.
  Interventions: Drug: Upadacitinib
- Study 2: Group 2 Upadacitinib Dose B (Experimental): Participants will receive upadacitinib Dose B once daily for 52 weeks in Period A and Period B.
  Interventions: Drug: Upadacitinib
- Study 2: Group 3 Placebo (Experimental): Participants will receive matching placebo once daily for 24 weeks in Period A.
  Interventions: Drug: Placebo
- Study 2: Group 4 Upadacitinib Dose A (Experimental): Participants initially randomized to placebo (Period A) with a SALT score > 20 at Week 24 will be re-randomized to receive upadacitinib Dose A once daily for 28 weeks in Period B.
  Interventions: Drug: Upadacitinib; Drug: Placebo
- Study 2: Group 5 Upadacitinib Dose B (Experimental): Participants initially randomized to placebo (Period A) with a SALT score > 20 at Week 24 will be re-randomized to receive upadacitinib Dose B once daily for 28 weeks in Period B.
  Interventions: Drug: Upadacitinib; Drug: Placebo
- Study 2: Group 6 Placebo (Experimental): Participants initially randomized to placebo with a SALT score ≤ 20 at Week 24 will continue on placebo through Week 160.
  Interventions: Drug: Placebo
- Study 3: Group 1 Upadacitinib Dose B (SALT > 20) (Experimental): Participants receiving upadacitinib Dose A with a SALT score > 20 at Week 52 (end of Period B) of Study 1 or Study 2 will dose escalate to upadacitinib Dose B once daily for 108 weeks.
  Interventions: Drug: Upadacitinib
- Study 3: Group 2 Upadacitinib Dose A (SALT ≤ 20) (Experimental): Participants receiving upadacitinib Dose A with a SALT score ≤ 20 at Week 52 (end of Period B) of Study 1 or Study 2 will remain on upadacitinib Dose A once daily for 108 weeks.
  Interventions: Drug: Upadacitinib
- Study 3: Group 3 Upadacitinib Dose B (Non-Sustained) (Experimental): Participants who end Period B on upadacitinib Dose B with a with a SALT score > 20 at Week 40 or Week 52 of Study 1 or Study 2 will remain on upadacitinib Dose B once daily for 108 weeks.
  Interventions: Drug: Upadacitinib
- Study 3: Group 4 Upadacitinib Dose B (Sustained) (Experimental): Participants who end Period B on upadacitinib Dose B with a with a SALT score ≤ 20 at Week 40 and Week 52 of Study 1 or Study 2 will be re-randomized to receive upadacitinib Dose B once daily for 108 weeks.
  Interventions: Drug: Upadacitinib
- Study 3: Group 5 Upadacitinib Dose A (Sustained) (Experimental): Participants who end Period B on upadacitinib Dose B with a with a SALT score ≤ 20 at Week 40 and Week 52 of Study 1 or Study 2 will be re-randomized to receive upadacitinib Dose A once daily for 108 weeks.
  Interventions: Drug: Upadacitinib
- Study 4: Group 1 Upadacitinib Dose A (Experimental): US only adolescent participants will receive upadacitinib Dose A once daily for 52 weeks in Period A and Period B.
  Interventions: Drug: Upadacitinib
- Study 4: Group 2 Upadacitinib Dose B (Experimental): US only adolescent participants will receive upadacitinib Dose B once daily for 52 weeks in Period A and Period B.
  Interventions: Drug: Upadacitinib
- Study 4: Group 3 Placebo (Experimental): US only adolescent participants will receive matching placebo once daily for 24 weeks in Period A.
  Interventions: Drug: Placebo
- Study 4: Group 4 Upadacitinib Dose A (Experimental): Participants initially randomized to placebo (Period A) with a SALT score > 20 at Week 24 will be re-randomized to receive upadacitinib Dose A once daily for 28 weeks in Period B.
  Interventions: Drug: Upadacitinib
- Study 4: Group 5 Upadacitinib Dose B (Experimental): Participants initially randomized to placebo (Period A) with a SALT score > 20 at Week 24 will be re-randomized to receive upadacitinib Dose B once daily for 28 weeks in Period B.
  Interventions: Drug: Upadacitinib
- Study 4: Group 6 Placebo (Experimental): Participants initially randomized to placebo with a SALT score ≤ 20 at Week 24 will continue on placebo through Week 160.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Upadacitinib — Oral Tablets
  Other Names: Rinvoq; ABT-494
  Arms: Study 1: Group 1 Upadacitinib Dose A; Study 1: Group 2 Upadacitinib Dose B; Study 1: Group 4 Upadacitinib Dose A; Study 1: Group 5 Upadacitinib Dose B; Study 2: Group 1 Upadacitinib Dose A; Study 2: Group 2 Upadacitinib Dose B; Study 2: Group 4 Upadacitinib Dose A; Study 2: Group 5 Upadacitinib Dose B; Study 3: Group 1 Upadacitinib Dose B (SALT > 20); Study 3: Group 2 Upadacitinib Dose A (SALT ≤ 20); Study 3: Group 3 Upadacitinib Dose B (Non-Sustained); Study 3: Group 4 Upadacitinib Dose B (Sustained); Study 3: Group 5 Upadacitinib Dose A (Sustained); Study 4: Group 1 Upadacitinib Dose A; Study 4: Group 2 Upadacitinib Dose B; Study 4: Group 4 Upadacitinib Dose A; Study 4: Group 5 Upadacitinib Dose B
Drug: Placebo — Oral Tablets
  Arms: Study 1: Group 3 Placebo; Study 1: Group 4 Upadacitinib Dose A; Study 1: Group 5 Upadacitinib Dose B; Study 1: Group 6 Placebo; Study 2: Group 3 Placebo; Study 2: Group 4 Upadacitinib Dose A; Study 2: Group 5 Upadacitinib Dose B; Study 2: Group 6 Placebo; Study 4: Group 3 Placebo; Study 4: Group 6 Placebo

SUMMARY:
Alopecia areata (AA) is a disease that happens when the immune system attacks hair follicles and causes hair loss. AA usually affects the head and face, but hair loss can happen on any part of the body. The purpose of this study is to assess how safe, effective, and tolerable upadacitinib is in adolescent and adult participants with severe AA.

Upadacitinib is an approved drug being investigated for the treatment of AA. In Study 1 and Study 2 and Study 4 Period A, participants are placed in 1 of 3 groups, called treatment arms. Each group receives a different treatment. There is a 1 in 5 chance that participants will be assigned to placebo. In Study 1 and Study 2 and Study 4 Period B, participants originally randomized to upadacitinib dose group in Period A will continue their same treatment in Period B. Participants originally randomized to Placebo in Period A will either remain on placebo in Period B, or be randomized in 1 of 2 groups, based off of their Severity of Alopecia Tool (SALT) score. Participants who complete Study 1, Study 2 or Study 4, can join Study 3 and may be re-randomized to receive 1 of 2 doses of upadacitinib for up to 108 weeks. Around 1500 participants with severe AA will be enrolled in the study at approximately 280 sites worldwide.

Participants will receive oral tablets of either upadacitinib or placebo once daily for up to 160 weeks with the potential of being re-randomized into a different treatment group at Weeks 24 and 52. Participants will be followed up for up to 30 days after last study drug dose.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Adult individuals must be < 64 years old at Baseline Visit. Where permitted outside United States (US)/European Union (EU), adolescent individuals who are at least 12 years old at Screening may participate in Study 1 and Study 2. Adolescent individuals in the US who are at least 12 years old at Screening may participate in Study 4.
* Diagnosis of severe alopecia areata (AA) with Severity of Alopecia Tool (SALT) score >= 50 scalp hair loss at Screening and Baseline.
* Severe AA with no spontaneous scalp hair regrowth over the past 6 months.
* Current episode of AA of less than 8 years.

Exclusion Criteria:

* Current diagnosis of primarily diffuse type of AA.
* Current diagnosis of other types of alopecia that would interfere with evaluation of AA, including but not limited to female pattern hair loss, male pattern hair loss (androgenetic alopecia) Stage III or greater based on Hamilton-Norwood classification, traction alopecia, lichen planopilaris (LPP), discoid lupus, frontal fibrosing alopecia (FFA), central centrifugal cicatricial alopecia (CCCA), folliculitis decalvans, trichotillomania, and telogen effluvium.
* Diagnosis of other types of inflammatory scalp, eyebrow, or eyelash disorders that would interfere with evaluation of AA as determined by the investigator, including but not limited to seborrheic dermatitis, scalp psoriasis, atopic dermatitis (AD), and tinea capitis.

Ages: 12 Years to 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1500 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with the Achievement of Severity of Alopecia Tool (SALT) Score <= 20 | Week 24
  The SALT is a global AA severity score based on the combination of extent and density of scalp hair loss. The score is determined by visually defining the amount of terminal hair loss in each of the 4 views of the scalp (left and right side each accounting for 18% of scalp area, the top for 40%, and the back for 24%) and adding these together with a maximum score of 100%.
Number of Participants with Adverse Events (AEs) | Up to approximately 164 weeks
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation in which a participant is administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Achievement of SALT score <= 20 for the Comparison of Upadacitinib Dose A QD Versus Placebo | Week 24
  The SALT is a global AA severity score based on the combination of extent and density of scalp hair loss. The score is determined by visually defining the amount of terminal hair loss in each of the 4 views of the scalp (left and right side each accounting for 18% of scalp area, the top for 40%, and the back for 24%) and adding these together with a maximum score of 100%.
Percentage of Participants with the Achievement of SALT Score <= 10 | Up to Week 24
  The SALT is a global AA severity score based on the combination of extent and density of scalp hair loss. The score is determined by visually defining the amount of terminal hair loss in each of the 4 views of the scalp (left and right side each accounting for 18% of scalp area, the top for 40%, and the back for 24%) and adding these together with a maximum score of 100%.
Percentage of Participants with the Achievement of SALT Score <= 20 | Up to Week 12
  The SALT is a global AA severity score based on the combination of extent and density of scalp hair loss. The score is determined by visually defining the amount of terminal hair loss in each of the 4 views of the scalp (left and right side each accounting for 18% of scalp area, the top for 40%, and the back for 24%) and adding these together with a maximum score of 100%.
Percentage of Participants with the Achievement of Clinician-Reported Outcome (ClinRO) Measure for Eyebrow Hair Loss of 0 or 1 | Baseline to Week 24
  The ClinRO for Eyebrow Hair Loss is a 4-point response scale where 0 = The eyebrows have full coverage and no areas of hair loss and 3 = No notable eyebrows. Responses should have a ≥ 2-point improvement from Baseline among participants with Baseline score ≥ 2.
Percentage of Participants with the Achievement of ClinRO Measure for Eyelash Hair Loss of 0 or 1 | Baseline to Week 24
  The ClinRO for Eyelash Hair Loss is a 4-point response scale where 0 = The eyelashes form a continuous line along the eyelids on both eyes and 3 = No notable eyelashes. Responses should have a ≥ 2-point improvement from Baseline among participants with Baseline score ≥ 2.
Percentage of Participants with the Achievement of SALT 75 | Baseline to Week 24
  SALT 75 is defined as at least a 75% improvement [decrease] from Baseline in SALT score.
Percentage of Participants with the Achievement of SALT 90 | Baseline to Week 24
  SALT 90 is defined as at least a 90% improvement [decrease] from Baseline in SALT score.
Percent Change from Baseline in SALT Score | Baseline to Week 24
  The SALT is a global AA severity score based on the combination of extent and density of scalp hair loss. The score is determined by visually defining the amount of terminal hair loss in each of the 4 views of the scalp (left and right side each accounting for 18% of scalp area, the top for 40%, and the back for 24%) and adding these together with a maximum score of 100%.
Percentage of Participants with the Achievement of Patients' Global Impression of Change of Alopecia Areata (PaGIC-AA) Score of 1 "Much Better" or 2 "Moderately Better" | Up to Week 24
  The PaGIC-AA is a single-item measure that asks participants to rate how their alopecia condition has changed overall since the start of the study using a 7-point scale. Responses range from "much better" to "much worse."
Percentage of Participants with the Achievement of Patient-Reported Outcome (PRO) for Scalp Hair Assessment 0/1 with ≥ 2-Point Improvement (Reduction) | Baseline to Week 24
  The PRO for Scalp Hair Assessment is single item, five-point, categorical response scale that asks respondents to look in the mirror and assess the total area of the scalp with missing hair. Response items range from "No missing hair" to "Nearly all or all" and includes percentage ranges for each category (0%, 1 to 20%, 21 to 49%, 50 to 94%, and 95 to 100%). Responses among participants with baseline score >=3.
Change from Baseline in Alopecia Areata Symptom Impact Scale (AASIS) Interference Subscale Score | Week 24
  The AASIS Interference Subscale is a 6-item assessment with scores ranging from 0 = 'did not interfere' to 10 = 'interfered completely' with higher scores indicating greater symptom interference.
Change from Baseline in AASIS Symptoms Subscale Score | Week 24
  The AASIS Symptom Subscale is a 7-item assessment with scores ranging from 0 = 'not present' to 10 = 'as bad as you can imagine' with higher scores indicating greater symptom severity.
Change from Baseline in Skindex-16 AA Emotions Domain Scores | Week 24
  The Skindex-16 AA Emotions Domain is a 7-item assessment ranging from 0 = never bothered to 6 = always bothered that measures the effects of AA on a subject's health-related quality of life. Higher scores indicate greater impact on health-related quality of life.
Change from Baseline in Skindex-16 AA Functioning Domain Scores | Week 24
  The Skindex-16 AA Emotions Domain is a 5-item assessment ranging from 0 = never bothered to 6 = always bothered, that measures the effects of AA on a subject's health-related quality of life. Higher scores indicate greater impact on health-related quality of life.
Achievement of Hospital Anxiety and Depression Scale (HADS)-Anxiety < 8 and HADS-Depression < 8 at Week 24 Among Participants with HADS-A >= 8 or HADS-D >= 8 at Baseline | Baseline to Week 24
  The HADS is a self-administered scale which measures anxiety and depression. It contains 14 items and is comprised of anxiety (7 items) and depression (7 items) subscales, which are scored separately and summed to give a total score. Item scores range from 0 (best) to 3 (worst), and total scores are categorized as normal (0 to 7), borderline abnormal (8 to 10), and abnormal (11 to 21).
Percentage of Participants with the Achievement of SALT Score 0 | Week 24
  The SALT is a global AA severity score based on the combination of extent and density of scalp hair loss. The score is determined by visually defining the amount of terminal hair loss in each of the 4 views of the scalp (left and right side each accounting for 18% of scalp area, the top for 40%, and the back for 24%) and adding these together with a maximum score of 100%.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (267):
- United States (73):
  - Total Skin and Beauty Dermatology Center /ID# 259539, Birmingham, Alabama
  - Duplicate_Advanced Research Associates - Glendale /ID# 259108, Glendale, Arizona
  - Southwest Skin Specialists /ID# 258234, Phoenix, Arizona
  - Alliance Dermatology and Mohs Center /ID# 258111, Phoenix, Arizona
  - Johnson Dermatology Clinic /ID# 259103, Fort Smith, Arkansas
  - Duplicate_JOSEPH RAOOF MD,INC /ID# 258031, Encino, California
  - First OC Dermatology /ID# 259220, Fountain Valley, California
  - University of California Irvine /ID# 259096, Irvine, California
  - Dermatology Research Associates /ID# 258033, Los Angeles, California
  - Stanford University School of Medicine - Redwood City /ID# 259542, Redwood City, California
  - Integrative Skin Science and Research /ID# 258114, Sacramento, California
  - University of California Davis Health /ID# 258112, Sacramento, California
  - Clinical Trials Research Institute /ID# 258021, Thousand Oaks, California
  - Skin Care Research Boca Raton /ID# 258012, Boca Raton, Florida
  - Apex Clinical Trials /ID# 259205, Brandon, Florida
  - Florida Academic Dermatology Center /ID# 259353, Coral Gables, Florida
  - Skin Research Institute LLC /ID# 259207, Coral Gables, Florida
  - Revival Research /ID# 259213, Doral, Florida
  - Skin Care Research - Hollywood /ID# 259210, Hollywood, Florida
  - GSI Clinical Research, LLC /ID# 259352, Margate, Florida
  - Life Clinical Trials /ID# 259358, Margate, Florida
  - Lenus Research and Medical Group /ID# 259356, Miami, Florida
  - International Clinical Research - Sanford /ID# 259547, Sanford, Florida
  - FWD Clinical Research /ID# 266687, Tamarac, Florida
  - Advanced Clinical Research Institute /ID# 259204, Tampa, Florida
  - Avita Clinical Research /ID# 258011, Tampa, Florida
  - Cleaver Medical Group Dermatology /ID# 259801, Dawsonville, Georgia
  - Marietta Dermatology /ID# 259818, Marietta, Georgia
  - Northwestern University Feinberg School of Medicine /ID# 259555, Chicago, Illinois
  - NorthShore University HealthSystem - Skokie /ID# 266684, Skokie, Illinois
  - Indiana University Health University Hospital /ID# 259827, Indianapolis, Indiana
  - U.S. Dermatology Partners Leawood /ID# 259203, Leawood, Kansas
  - Tulane University School of Medicine /ID# 259799, New Orleans, Louisiana
  - Raven Clinical Research /ID# 268453, Marriottsville, Maryland
  - MetroBoston Clinical Partners /ID# 259559, Boston, Massachusetts
  - Lahey Hospital & Medical Center /ID# 260484, Burlington, Massachusetts
  - Great Lakes Research Group - Bay City /ID# 259100, Bay City, Michigan
  - Hamzavi Dermatology - Canton /ID# 260115, Canton, Michigan
  - Clin Res Inst of Michigan, LLC /ID# 259802, Chesterfield, Michigan
  - Clarkston Dermatology /ID# 258018, Clarkston, Michigan
  - Henry Ford Medical Center - New Center One /ID# 258067, Detroit, Michigan
  - M Health Fairview University of Minnesota Medical Center - East Bank /ID# 260122, Minneapolis, Minnesota
  - Minnesota Clinical Study Center /ID# 259218, New Brighton, Minnesota
  - Dermatology and Skin Center of Lees Summit /ID# 259206, Lee's Summit, Missouri
  - Physician Research Collaboration, LLC /ID# 259354, Lincoln, Nebraska
  - Skin Specialists /ID# 259237, Omaha, Nebraska
  - Skin Cancer and Dermatology Institute - Reno /ID# 259208, Reno, Nevada
  - The Skin Center Dermatology Group /ID# 266748, New City, New York
  - Schweiger Dermatology, P.C. /ID# 258007, New York, New York
  - Schweiger Dermatology, P.C. /ID# 259531, New York, New York
  - Equity Medical, LLC /ID# 266680, New York, New York
  - Icahn School of Medicine at Mount Sinai /ID# 259808, New York, New York
  - Sadick Research Group LLC /ID# 266790, New York, New York
  - Piedmont Plastic Surgery and Dermatology /ID# 258206, Huntersville, North Carolina
  - Cleveland Clinic - Cleveland /ID# 258113, Cleveland, Ohio
  - Remington-Davis Clinical Research /ID# 258106, Columbus, Ohio
  - Dermatologists of Southwest Ohio, Inc /ID# 260116, Mason, Ohio
  - Dermatologist of Central States (DOCS) Clinical Research - Springfield /ID# 266746, Springfield, Ohio
  - Oregon Dermatology and Research Center /ID# 258243, Portland, Oregon
  - Oregon Medical Research Center /ID# 258107, Portland, Oregon
  - University of Pittsburgh Medical Center /ID# 266681, Pittsburgh, Pennsylvania
  - Medical University of South Carolina /ID# 259828, Charleston, South Carolina
  - Health Concepts /ID# 266678, Rapid City, South Dakota
  - International Clinical Research - Tennessee LLC /ID# 259552, Murfreesboro, Tennessee
  - Arlington Research Center, Inc /ID# 258028, Arlington, Texas
  - Bellaire Dermatology Associates /ID# 259360, Bellaire, Texas
  - U.S. Dermatology Partners - Cedar Park /ID# 259367, Cedar Park, Texas
  - Dermatology Treatment and Research Center /ID# 259357, Dallas, Texas
  - Modern Research Associates, PLLC /ID# 259349, Dallas, Texas
  - Reveal Research Institute - Dallas /ID# 259361, Dallas, Texas
  - Center for Clinical Studies - Houston - Northwest Freeway /ID# 258036, Houston, Texas
  - Progressive Clinical Research /ID# 259365, San Antonio, Texas
  - Complete Dermatology /ID# 258025, Sugar Land, Texas
- Argentina (5):
  - Buenos Aires Skin /ID# 258297, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Instituto de Neumonologia y Dermatologia /ID# 258640, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Psoriahue Med Interdisciplinar /ID# 258641, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Instituto De Investigaciones Clínicas Córdoba /ID# 260244, Córdoba, Córdoba Province
  - Centro de Investigacion y Prevencion Cardiovascular (CIPREC) /ID# 258639, Buenos Aires
- Australia (8):
  - Momentum Clinical Research /ID# 258571, Darlinghurst, New South Wales
  - St George Dermatology & Skin Cancer Centre /ID# 258567, Kogarah, New South Wales
  - Cornerstone Dermatology /ID# 258769, Coorparoo, Queensland
  - Veracity Clinical Research /ID# 258566, Woolloongabba, Queensland
  - Skin Health Institute Inc /ID# 258570, Carlton, Victoria
  - Sinclair Dermatology - Melbourne /ID# 258565, East Melbourne, Victoria
  - The Royal Melbourne Hospital /ID# 258770, Parkville, Victoria
  - Fremantle Dermatology /ID# 260207, Fremantle, Western Australia
- Belgium (6):
  - Universite Libre de Bruxelles - Hopital Erasme /ID# 257314, Anderlecht, Brussels Capital
  - Cliniques Universitaires UCL Saint-Luc /ID# 257320, Brussels, Brussels Capital
  - Universitair Ziekenhuis Brussel /ID# 257325, Jette, Brussels Capital
  - UZ Gent /ID# 257317, Ghent, Oost-Vlaanderen
  - AZ Delta - campus Torhout /ID# 257321, Torhout, West-Vlaanderen
  - CHU de Liege /ID# 257316, Liège
- Brazil (5):
  - Irmandade da Santa Casa de Misericordia de Porto Alegre /ID# 258045, Porto Alegre, Rio Grande do Sul
  - Upeclin Fmb - Unesp /Id# 258046, Botucatu, São Paulo
  - Hospital e Maternidade Celso Pierro - PUC-Campinas /ID# 258105, Campinas, São Paulo
  - Instituto Brasil de Pesquisa Clinica S.A - IBPClin /ID# 258750, Rio de Janeiro
  - Hospital Alemao Oswaldo Cruz /ID# 258104, São Paulo
- Bulgaria (6):
  - Diagnostic Consultative Center Aleksandrovska /ID# 257049, Sofiya, Sofia
  - Diagnostic Consultative Centre (Dcc) - Foкus 5 /ID# 257048, Sofiya, Sofia
  - Diagnosis - Consult Centre 20 - Sofia /ID# 257273, Sofiya, Sofia
  - UMHAT Sveti Georgi /ID# 257548, Plovdiv
  - Duplicate_Ambulatory for Specialized Medical Care-IPSMC-skin and venereal diseas /ID# 257047, Sofia
  - UMHAT Professor Stoyan Kirkovich /ID# 257051, Stara Zagora
- Canada (16):
  - Dermatology Research Institute - Blackfoot Trail /ID# 258818, Calgary, Alberta
  - Beacon Dermatology Inc /ID# 258817, Calgary, Alberta
  - Rejuvenation Dermatology - Edmonton Downtown /ID# 258816, Edmonton, Alberta
  - Dr. Chih-ho Hong Medical Inc. /ID# 258814, Surrey, British Columbia
  - Wiseman Dermatology Research /ID# 258819, Winnipeg, Manitoba
  - SimcoDerm Medical and Surgical Dermatology Center /ID# 258820, Barrie, Ontario
  - Medicor Research Inc /ID# 258810, Greater Sudbury, Ontario
  - Leader Research /ID# 267028, Hamilton, Ontario
  - Lynderm Research Inc /ID# 258815, Markham, Ontario
  - JRB Research /ID# 259248, Ottawa, Ontario
  - SKiN Centre for Dermatology /ID# 258813, Peterborough, Ontario
  - York Dermatology Clinic & Research Centre /ID# 267026, Richmond Hill, Ontario
  - Private Practice - Dr. Kim Papp Clinical Research /ID# 259249, Waterloo, Ontario
  - Innovaderm Research Inc. /ID# 258812, Montreal, Quebec
  - Centre de Recherche dermatologique du Quebec Metropolitain /ID# 258811, Québec, Quebec
  - Private Practice - Dr. Angelique Gagne-Henley /ID# 267027, Saint-Jérôme, Quebec
- Chile (4):
  - Centro Medico Skin Med SPA /ID# 259314, Las Condes, Region Metropolitana Santiago
  - Centro Internacional de Estudios Clinicos - CIEC /ID# 259312, Santiago, Region Metropolitana Santiago
  - Clinica Dermacross /ID# 259311, Vitacura, Region Metropolitana Santiago
  - Fundacion Innovacion Cardiovascular /ID# 259313, Independencia, Santiago Metropolitan
- China (25):
  - Beijing Chaoyang Hospital,Capital Medical University /ID# 258912, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital /ID# 258941, Beijing, Beijing Municipality
  - Peking University People's Hospital /ID# 258940, Beijing, Beijing Municipality
  - Beijing Tongren Hospital Affiliated To Capital Medical University /ID# 266715, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University /ID# 260254, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital, Sun Yat-sen University /ID# 257367, Guangzhou, Guangdong
  - Dermatology Hospital of Southern Medical University /ID# 257118, Guangzhou, Guangdong
  - The First Affiliated Hospital Of Guangzhou Medical University /ID# 258663, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University /ID# 258485, Guangzhou, Guangdong
  - Shenzhen People's Hospital /ID# 258208, Shenzhen, Guangdong
  - Shenzhen Second Peoples Hospital /ID# 258060, Shenzhen, Guangdong
  - Union Hospital - Tongji Medical College /ID# 266737, Wuhan, Hubei
  - Renmin Hospital of Wuhan University /ID# 260260, Wuhan, Hubei
  - Dermatology Hospital of Jiangxi Provincial /ID# 259488, Nanchang, Jiangxi
  - The First Hospital of Jilin University /ID# 257496, Changchun, Jilin
  - Second Affiliated Hospital of Xian Jiaotong University /ID# 257497, Xi'an, Shaanxi
  - Shandong Dermatological Hospital /ID# 267520, Jinan, Shandong
  - Huashan Hospital, Fudan University /ID# 257758, Shanghai, Shanghai Municipality
  - First Affiliated Hospital of Shanxi Medical University /ID# 259647, Taiyuan, Shanxi
  - Chengdu Second Municipal People's Hospital /ID# 259492, Chengdu, Sichuan
  - West China Hospital, Sichuan University /ID# 259560, Chengdu, Sichuan
  - Tianjin Medical University General Hospital /ID# 259525, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine /ID# 257260, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine /ID# 257119, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University /ID# 257739, Wenzhou, Zhejiang
- Croatia (5):
  - DermaPlus - Poliklinika za dermatologiju i venerologiju /ID# 257151, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Zagreb /ID# 257630, Zagreb, City of Zagreb
  - Poliklinika Solmed /ID# 257651, Zagreb, City of Zagreb
  - Specialty Hospital Medico /ID# 257629, Rijeka, Primorje-Gorski Kotar County
  - Klinicki Bolnicki Centar (KBC) Split /ID# 257632, Split, Split-Dalmatia County
- France (10):
  - Chu de Nice-Hopital Larchet Ii /Id# 256978, Nice, Alpes-Maritimes
  - Hopital Ponchaillou /ID# 257520, Rennes, Brittany Region
  - Centre Hospitalier Universitaire de Bordeaux - Groupe Hospitalier Saint-Andre /ID# 257519, Bordeaux, Gironde
  - CHU Toulouse - Hopital Larrey /ID# 256980, Toulouse, Haute-Garonne
  - Polyclinique Courlancy /ID# 256977, Reims, Marne
  - Centre Hospitalier Universitaire de Nantes, Hotel Dieu -HME /ID# 256982, Nantes, Pays de la Loire Region
  - HCL - Hopital Edouard Herriot /ID# 256983, Lyon, Rhone
  - CHRU de Brest - Hopital Morvan /ID# 256979, Brest
  - Centre de Sante Sabouraud /ID# 257213, Paris
  - Hôpital Charles-Nicolle /ID# 256981, Rouen
- Germany (6):
  - TUM Klinikum rechts der Isar /ID# 257609, Munich, Bavaria
  - Fachklinik Bad Bentheim /ID# 257741, Bad Bentheim, Lower Saxony
  - Universitaetsklinikum Duesseldorf /ID# 257307, Düsseldorf, North Rhine-Westphalia
  - Universitaetsklinikum Muenster /ID# 257306, Münster, North Rhine-Westphalia
  - Universitaetsklinikum Schleswig-Holstein Campus Luebeck /ID# 257305, Lübeck, Schleswig-Holstein
  - Charite Universitaetsmedizin Berlin - Campus Mitte /ID# 257310, Berlin
- Greece (4):
  - General Hospital Andreas Syggros /ID# 257259, Athens, Attica
  - General Hospital Andreas Syggros /ID# 257262, Athens, Attica
  - Hospital of Skin and Venereal Diseases- Thessaloniki /ID# 257263, Thessaloniki
  - Papageorgiou General Hospital /ID# 257258, Thessaloniki
- Hungary (6):
  - Pecsi Tudomanyegyetem Klinikai Kozpont /ID# 257468, Pécs, Baranya
  - Bacs-Kiskun Varmegyei Oktatokorhaz /ID# 257472, Kecskemét, Bács-Kiskun county
  - Bagoly Egeszseghaz (Meditres Kft.) /ID# 258032, Kecskemét, Bács-Kiskun county
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont /ID# 258552, Szeged, Csongrád megye
  - Debreceni Egyetem-Klinikai Kozpont /ID# 257465, Debrecen, Hajdú-Bihar
  - DERMA-B Egeszsegugyi es Szolgaltato - Debrecen - Gyepusor Utca /ID# 257469, Debrecen
- Israel (5):
  - Hadassah Medical Center-Hebrew University /ID# 257946, Jerusalem, Jerusalem
  - The Chaim Sheba Medical Center /ID# 257770, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 257771, Tel Aviv, Tel Aviv
  - Rambam Health Care Campus /ID# 257769, Haifa
  - Rabin Medical Center. /ID# 257772, Petah Tikva
- Italy (12):
  - AZIENDA USL TOSCANA CENTRO - Ospedale Piero Palagi /ID# 257501, Florence, Firenze
  - ASL 1 Abruzzo - Ospedale regionale San Salvatore /ID# 257506, L’Aquila, L Aquila
  - IRCCS Istituto Clinico Humanitas /ID# 257500, Rozzano, Lombardy
  - Azienda Ospedaliera Universitaria Federico II /ID# 257504, Naples, Napoli
  - Azienda Ospedaliera Universitaria Luigi Vanvitelli /ID# 258585, Naples, Napoli
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata /ID# 257502, Rome, Roma
  - Azienda Ospedaliero-Universitaria Policlinico Umberto I /ID# 257513, Rome, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Universita Cattolica /ID# 257505, Rome, Roma
  - IRCCS AOU di Bologna Policlinico Sant Orsola Malpighi /ID# 257499, Bologna
  - ASST degli Spedali Civili di Brescia /ID# 257508, Brescia
  - AOU Policlinico G. Rodolico - San Marco /ID# 257507, Catania
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico /ID# 257503, Milan
- Japan (8):
  - Kurume University Hospital /ID# 257255, Kurume-shi, Fukuoka
  - Kitasato University Hospital /ID# 257285, Sagamihara-shi, Kanagawa
  - Niigata University Medical & Dental Hospital /ID# 259425, Niigata, Niigata
  - Osaka Metropolitan University Hospital /ID# 257256, Osaka, Osaka
  - Hamamatsu University Hospital /ID# 257253, Hamamatsu, Shizuoka
  - Kyorin University Hospital /ID# 257283, Mitaka-shi, Tokyo
  - Tokyo Medical University Hospital /ID# 258132, Shinjuku-ku, Tokyo
  - Yamaguchi University Hospital /ID# 257252, Ube-shi, Yamaguchi
- New Zealand (4):
  - Greenlane Clinical Centre /ID# 258563, Epsom, Auckland
  - Clinical Trials New Zealand /ID# 258564, Hamilton, Waikato Region
  - Aotearoa Clinical Trials /ID# 258562, Auckland
  - P3 Research Ltd /ID# 259846, Wellington
- Poland (10):
  - Dermodent Centrum Medyczne Aldona Czajkowska Rafał Czajkowski /ID# 258242, Osielsko, Kuyavian-Pomeranian Voivodeship
  - MICS Centrum Medyczne Torun / Nasz Lekarz Przychodnie Medyczne /ID# 257740, Torun, Kuyavian-Pomeranian Voivodeship
  - Specjalistyczny Gabinet Dermatologiczny Aplikacyjno Badawczy /ID# 257534, Krakow, Lesser Poland Voivodeship
  - Klinika Osipowicz & Turkowski sp.z.o.o /ID# 257598, Warsaw, Masovian Voivodeship
  - Royalderm Agnieszka Nawrocka /ID# 257536, Warsaw, Masovian Voivodeship
  - Osteo Medic s.c. Artur Racewicz Jerzy Supronik /ID# 257531, Bialystok, Podlaskie Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o. /ID# 257535, Gdansk, Pomeranian Voivodeship
  - Centrum Medyczne Angelius Provita /ID# 257916, Katowice, Silesian Voivodeship
  - Centrum Kliniczno-Badawcze J.Brzezicki, B. Gornikiewicz-Brzezicka Lekarze Spolka /ID# 257537, Elblag, Warmian-Masurian Voivodeship
  - Centrum Medyczne ALL-MED Badania Kliniczne /ID# 257590, Krakow
- Portugal (3):
  - Unidade Local de Saude de Almada-Seixal, EPE /ID# 257425, Almada, Setúbal District
  - Hospital CUF Descobertas /ID# 257419, Lisbon
  - Unidade Local de Saude de Santo Antonio, E.P.E. /ID# 258554, Porto
- Puerto Rico (5):
  - Santa Cruz Behavioral (SCB) Research Center /ID# 259350, Bayamón
  - Dr. Samuel Sanchez PSC /ID# 259359, Caguas
  - Clinical Research Puerto Rico /ID# 259355, San Juan
  - GCM Medical Group PSC /ID# 258013, San Juan
  - Mindful Medical Research /ID# 260113, San Juan
- Slovakia (4):
  - Univerzitna nemocnica Bratislava, Nemocnica Stare mesto /ID# 257594, Bratislava, Bratislava Region
  - Derma therapy spol /ID# 257595, Bratislava, Bratislava Region
  - Fakultna nemocnica s poliklinikou J.A. Reimana Presov /ID# 257593, Prešov, Presov
  - Kaderma Majtan s.r.o. /ID# 257596, Topoľčany
- South Korea (11):
  - Pusan National University Hospital /ID# 257910, Busan, Busan Gwang Yeogsi
  - Kyungpook National University Hospital /ID# 257908, Daegu, Daegu Gwang Yeogsi
  - Chungnam National University Hospital /ID# 267151, Daejeon, Daejeon Gwang Yeogsi
  - Seoul National University Bundang Hospital /ID# 257906, Seongnam-si, Gyeonggido
  - Inha University Hospital /ID# 257904, Incheon, Incheon Gwang Yeogsi
  - Jeonbuk National University Hospital /ID# 267154, Jeonju, Jeonrabugdo
  - Chungang University Hospital /ID# 267155, Dongjak-gu, Seoul Teugbyeolsi
  - Seoul National University Hospital /ID# 257903, Seoul, Seoul Teugbyeolsi
  - Konkuk University Medical Center /ID# 257900, Seoul, Seoul Teugbyeolsi
  - Kyung Hee University Hospital at Gangdong /ID# 257907, Seoul, Seoul Teugbyeolsi
  - Hallym University Kangdong Sacred Heart Hospital /ID# 257905, Seoul
- Spain (6):
  - Hospital Universitari de Bellvitge /ID# 257332, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Reina Sofia /ID# 257035, Córdoba, Cordoba
  - Hospital Universitario de Fuenlabrada /ID# 257334, Fuenlabrada, Madrid
  - Hospital Santa Creu i Sant Pau /ID# 257034, Barcelona
  - Hospital Universitario La Paz /ID# 257333, Madrid
  - Hospital Universitario Dr. Peset /ID# 257036, Valencia
- Sweden (3):
  - Karolinska University Hospital Solna /ID# 257094, Solna, Stockholm County
  - Diagnostiskt Centrum Hud /ID# 257229, Stockholm, Stockholm County
  - CTC GoCo /ID# 257714, Mölndal, Västra Götaland County
- Taiwan (5):
  - Kaohsiung Chang Gung Memorial Hospital /ID# 258726, Kaohsiung City, Kaohsiung
  - National Taiwan University Hospital /ID# 257407, Taipei City, Taipei
  - National Cheng Kung University Hospital /ID# 257409, Tainan
  - Taipei Veterans General Hosp /ID# 257413, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 258725, Taoyuan
- Turkey (Türkiye) (5):
  - Gulhane Egitim ve Arastirma Hastanesi /ID# 257509, Ankara, Antalya
  - Ankara City Hospital /ID# 257417, Ankara
  - Gaziantep Universitesi /ID# 257418, Gaziantep
  - Bagcilar Medipol Mega Universite Hastanesi /ID# 257449, Istanbul
  - Erciyes University Medical Faculty /ID# 259034, Kayseri
- United Kingdom (7):
  - Velocity Clinical Research Ltd /ID# 257925, High Wycombe, Buckinghamshire
  - Royal Sussex County Hospital /ID# 257912, Brighton, East Sussex
  - Gloucestershire Royal Hospital /ID# 257953, Gloucester, Gloucestershire
  - Chelsea and Westminster Hospital /ID# 259128, London, Greater London
  - Oxford University Hospitals NHS Foundation Trust /ID# 257948, Oxford, Oxfordshire
  - London North West University Healthcare NHS Trust /ID# 257914, Harrow
  - Northern Care Alliance NHS Group /ID# 257952, Salford

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M23-716